CLINICAL TRIAL: NCT05159349
Title: Mental Health During the Whole Life Cycle of Community Patients with Schizophrenia: a Cohort Study
Brief Title: Mental Health During the Whole Life Cycle of Community Patients with Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: Jun-Cai
Record Dates: First submitted 2021-11-10; First posted 2021-12-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cohort study; The whole life cycle; Mental health
MeSH Terms: conditions — Schizophrenia; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Proteomics: collecting peripheral blood(5ml), once a year.
  2. Genomics: collecting peripheral blood( 2ml), collected at enrollment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed group
- Non-exposed group

SUMMARY:
Schizophrenia is one of the components of severe mental disorders. It has the characteristics of prolonged course, low cure rate, high recurrence rate and high disability rate. It brings many short-term and long-term effects to individuals, families and society. Studies on patients with schizophrenia mainly focus on cross-sectional and case-control studies, but there is a lack of long-term follow-up of patients with schizophrenia in the community. Therefore, this study would establish a cohort study to solve the chronological relationship between exposure and effect, focus on community schizophrenia, and establish a community schizophrenia patient biobank that has been tracked for a long time from diagnosis.

DETAILED DESCRIPTION:
Schizophrenia is one of the components of severe mental disorders. It has the characteristics of prolonged course, low cure rate, high recurrence rate and high disability rate. It brings many short-term and long-term effects to individuals, families and society.Studies on patients with schizophrenia mainly focus on cross-sectional and case-control studies, but there is a lack of long-term follow-up of patients with schizophrenia in the community. Therefore, this study would establish a cohort study to solve the chronological relationship between exposure and effect, focus on community schizophrenia, and establish a community schizophrenia patient biobank that has been tracked for a long time from diagnosis.

1. Aim of the study:

   1.1 Based on previous studies, this study will focus on patients with schizophrenia in the community. Establishing a biobank of new cases to monitor the occurrence of disease recurrences, violent behaviours and other outcome events during the whole life cycle of schizophrenia patients. Exploring the predictive effects of biological, psychosocial, imaging and other indicators on patient recurrence and other events.

   1.2 At the same time, establishing a sample database of patients with schizophrenia in the community to lay a working foundation and reserve sample resources for subsequent related mechanism research, drug research, and intervention research.
2. Content of the study 2.1 At least 1,200 patients with schizophrenia diagnosed within five years will be recruited. On the basis of community follow-up and health examination, this study will expand biological sample collection and professional scale evaluation, establish a schizophrenia community cohort.

   2.2 Based on the establishment of the cohort, this study will carry out statistical description according to the type of data. The differences will be compared between the exposed group and the unexposed group in demographic information, family and past disease history, personal living habits, condition and treatment, psychological evaluation, social support evaluation, sleep quality, functional evaluation, quality of life and other content. Repeated measures analysis of variance will be used to compare the differences in blood pressure, blood glucose and other indicators between the exposed group and the unexposed group. The generalized estimating equation will be used to analyze the relationship between the outcome of recurrence and emergency about physical activity, related biochemical indicators, and social support. On the basis of statistical results, this study will carry out research on the prognostic factors and related physiological mechanisms of schizophrenia.
3. Study design 3.1 Pay attention to multiple prognostic outcomes such as relapse, dangerous behaviours, suicide and self-harm, calculate the included sample size based on this. After the start of the project, in Hongkou, Jinshan, Minhang, and Xuhui districts, all schizophrenic patients in management who meet the inclusion criteria will be continuously included in the district.

3.2 At baseline, the patient's demographic information and a complete health history (include personal history, family history, and medical history) will be taken. The questionnaire survey includes the Brief Psychiatric Rating Scale (BPRS)，the Patient Health Questionnaire-9 (PHQ-9)，the Generalized Anxiety Disorder Screener (GAD-7), the Pittsburgh Sleep Quality Index (PSQI) , the WHO Quality of Life Scale-Brief (WHOQOL-BREF) , the Modified Overt Aggression Scale (MOAS), the 10-item social disability screening schedule (SDSS) and the Perceived social support scale(PSSS),etc. Within six months of the completion of the baseline survey, the district-level mental health center arranges for patients in the district to participate in physical examinations. All measures will be administered at baseline and 12, 24, 36 and 48 months follow-up except for the health history and PSSS, which will be administered only at baseline. Besides, the study will focus on the patients' recurrence events, violent behavior, various impacts on society and family, emergency response events, and prognosis by carrying out active follow-up every three months.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Shanghai Mental Health Information Management System.
* Meets criteria for the diagnosis of schizophrenia (ICD-10 or ICD-11).
* Patients with schizophrenia diagnosed within five years.
* Age 18 years or older.

Exclusion Criteria:

* Patients with severe physical diseases and organic brain diseases.
* The patient is about to settle outside Shanghai.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since the start of the project, all schizophrenia patients in management who meet the inclusion criteria in this district have been continuously included in Hongkou, Jinshan, Minhang, and Xuhui districts, and at least 300 patients in each district will be included until the corresponding sample size is reached.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
1-year BPRS reduction rate | Change from Baseline BPRS at 12 months
  The Brief Psychiatric Rating Scale (BPRS) was used to measure the presence and severity of psychiatric symptoms entailing positive symptoms, general psychopathology, and affective symptoms (e.g., thought disturbance, emotional withdrawal, hostility, and suspiciousness) for patients with mental illness, particularly schizophrenia. Each of the 18 items are designed to represent a discrete symptom area. Items are rated on a 7-point Likert scale, from 1 = "not present" to 7 = "extremely severe", with scores ranging from 18 to 126 (achieved through summing the item scores). Higher scores indicated more severity of psychiatric symptoms.
  Reduction rate was calculated using the following formula: reduction rate= (Score before treatment - Score after treatment)/(Score before treatment - 18) × 100%. A reduction rate of BPRS score > 25% was considered as a clinically meaningful improvement.
2-year BPRS reduction rate | Change from Baseline BPRS at 24 months
  The BPRS reduction rate during the 2-year follow-up period.
3-year BPRS reduction rate | Change from Baseline BPRS at 36 months
  The BPRS reduction rate during the 3-year follow-up period.
4-year BPRS reduction rate | Change from Baseline BPRS at 48 months
  The BPRS reduction rate during the 4-year follow-up period.

SECONDARY OUTCOMES:
1-year MOAS | Change from Baseline MOAS at 12 months
  The Modified Overt Aggression Scale (MOAS) is a four-part behavior rating scale used to evaluate and document the "frequency and severity" of aggressive episodes. The rating scale is made up of four categories; verbal aggression, aggression against objects, aggression against self, and aggression against others. Each category consists of five responses, which over time can track the patient's aggressive behavior. The MOAS is one of the most widely used measures for violence and aggression, with 4 items in total, 0~4 points for each item.
2-year MOAS | Change from Baseline MOAS at 24 months
  The change in MOAS scores from baseline during the 2-year follow-up period.
3-year MOAS | Change from Baseline MOAS at 36 months
  The change in MOAS scores from baseline during the 3-year follow-up period.
4-year MOAS | Change from Baseline MOAS at 48 months
  The change in MOAS scores from baseline during the 4-year follow-up period.
1-year WHOQOL-BREF | Change from Baseline WHOQOL-BREF at 12 months
  The WHO Quality of Life Scale-Brief (WHOQOL-BREF) was developed by the Word Health Organisation as a quality of life assessment that would be applicable cross-culturally. It is a 26 item self report measure, especially useful for measuring outcomes with adults with a psychosocial disability. The WHOQOL-BREF measures four factors: physical health, psychological Health, social relationships, and environment. The total score is presented between 26 and 156, where higher scores represent higher levels of quality of life.
2-year WHOQOL-BREF | Change from Baseline WHOQOL-BREF at 24 months
  The change in WHOQOL-BREF scores from baseline during the 2-year follow-up period.
3-year WHOQOL-BREF | Change from Baseline WHOQOL-BREF at 36 months
  The change in WHOQOL-BREF scores from baseline during the 3-year follow-up period.
4-year WHOQOL-BREF | Change from Baseline WHOQOL-BREF at 48 months
  The change in WHOQOL-BREF scores from baseline during the 4-year follow-up period.
1-year GAD-7 | Change from Baseline GAD-7 at 12 months
  The Generalized Anxiety Disorder Screener (GAD-7) is a brief, 7-item self-report measure for anxiety symptoms in adolescents and adults. Although developed primarily as a screening tool for GAD, it can also be used as a diagnostic tool to monitor changes in symptoms over time, and as a screener for social anxiety, panic disorder, and post-traumatic stress disorder. Each item is rated on a likert-type scale from zero ("not at all") to three ("nearly every day"), with total scores ranging from 0 to 21.
2-year GAD-7 | Change from Baseline GAD-7 at 24 months
  The change in GAD-7 scores from baseline during the 2-year follow-up period.
3-year GAD-7 | Change from Baseline GAD-7 at 36 months
  The change in GAD-7 scores from baseline during the 3-year follow-up period.
4-year GAD-7 | Change from Baseline GAD-7 at 48 months
  The change in GAD-7 scores from baseline during the 4-year follow-up period.
1-year PHQ-9 | Change from Baseline PHQ-9 at 12 months
  The Patient Health Questionnaire-9 (PHQ-9) is a multipurpose instrument for screening , diagnosing , monitoring and measuring the severity of depression. The tool rates the frequency of the symptoms which factors into the scoring severity index. The PHQ -9 is brief and useful in clinical practice. The PHQ -9 can be administered repeatedly , which can reflect improvement or worsening of depression in response to treatment .Each item is rated on a likert-type scale from zero ("not at all") to three ("nearly every day").
2-year PHQ-9 | Change from Baseline PHQ-9 at 24 months
  The change in PHQ-9 scores from baseline during the 2-year follow-up period.
3-year PHQ-9 | Change from Baseline PHQ-9 at 36 months
  The change in PHQ-9 scores from baseline during the 3-year follow-up period.
4-year PHQ-9 | Change from Baseline PHQ-9 at 48 months
  The change in PHQ-9 scores from baseline during the 4-year follow-up period.
1-year PSQI | Change from Baseline PSQI at 12 months
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. The questionnaire consists of a combination of Likert- type and open-ended questions. Respondents are asked to indicate how frequently they have experienced certain sleep difficulties over the past month and to rate their overall sleep quality. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances.
2-year PSQI | Change from Baseline PSQI at 24 months
  The change in PSQI scores from baseline during the 2-year follow-up period.
3-year PSQI | Change from Baseline PSQI at 36 months
  The change in PSQI scores from baseline during the 3-year follow-up period.
4-year PSQI | Change from Baseline PSQI at 48 months
  The change in PSQI scores from baseline during the 4-year follow-up period.
1-year SDSS | Change from Baseline SDSS at 12 months
  The 10-item social disability screening schedule (SDSS) was used for measuring social function. It is a shortened version of psychiatric disability assessment schedule (DAS). SDSS was used to evaluate social disability, with 10 items in total, 0~2 points for each item.
2-year SDSS | Change from Baseline SDSS at 24 months
  The change in SDSS scores from baseline during the 2-year follow-up period.
3-year SDSS | Change from Baseline SDSS at 36 months
  The change in SDSS scores from baseline during the 3-year follow-up period.
4-year SDSS | Change from Baseline SDSS at 48 months
  The change in SDSS scores from baseline during the 4-year follow-up period.

OTHER OUTCOMES:
1-year Rate of rehospitalization | The rehospitalization rate from Baseline during the 1-year follow-up period.
  Relapse of patients with schizophrenia is defined as a clinical deterioration or an exacerbation of symptoms based on rehospitalization. Data from the Shanghai Mental Health Work Website.
2-year Rate of rehospitalization | From Baseline during the 2-year follow-up period.
  The rehospitalization rate from Baseline during the 2-year follow-up period.
3-year Rate of rehospitalization | From Baseline during the 3-year follow-up period.
  The rehospitalization rate from Baseline during the 3-year follow-up period.
4-year Rate of rehospitalization | From Baseline during the 4-year follow-up period.
  The rehospitalization rate from Baseline during the 4-year follow-up period.
1-year the number of violent incidents | From Baseline during the 1-year follow-up period.
  The primary health provider will follow up the patients every 3 months. If they learn about the violent behavior of the patient with schizophrenia during the follow-up process, they will record them on the Shanghai Mental Health Work Website.
2-year the number of violent incidents | From Baseline during the 2-year follow-up period.
  2-year the number of violent incidents
3-year the number of violent incidents | From Baseline during the 3-year follow-up period.
  3-year the number of violent incidents
4-year the number of violent incidents | From Baseline during the 4-year follow-up period.
  4-year the number of violent incidents
1-year the number of suicides | From Baseline during the 1-year follow-up period.
  The primary health provider will follow up the patients every 3 months. If they learn about the suicide in individuals with schizophrenia during the follow-up process, they will record them on the Shanghai Mental Health Work Website.
2-year the number of suicides | From Baseline during the 2-year follow-up period.
  2-year the number of suicides
3-year the number of suicides | From Baseline during the 3-year follow-up period.
  3-year the number of suicides
4-year the number of suicides | From Baseline during the 4-year follow-up period.
  4-year the number of suicides

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No